CLINICAL TRIAL: NCT01275248
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of Low-Dose Ondansetron For Adjunctive Therapy In Adult Patients With Obsessive-Compulsive Disorder Who Have Not Adequately Responded To Treatment With A Serotonin Reuptake Inhibitor
Brief Title: Efficacy and Safety Study of Low-Dose Ondansetron For Adjunctive Therapy In Adult Patients With Obsessive-Compulsive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Transcept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OND-003
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Obsessive-compulsive Disorder
Keywords: OCD; Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ondansetron 0.5 mg (Experimental): Ondansetron oral tablet 0.5 mg taken twice a day in addition to a serotonin reuptake inhibitor (SRI) for 12 weeks in the core period and for up to 30 months in the extension period.
  Interventions: Drug: Ondansetron
- Ondansetron 0.75 mg (Experimental): Ondansetron oral tablet 0.75 mg taken twice a day in addition to a serotonin reuptake inhibitor (SRI) for 12 weeks in the core period and for up to 30 months in the extension period.
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo oral tablet taken twice a day in addition to a serotonin reuptake inhibitor (SRI) for 12 weeks in the core period and for up to 30 months in the extension period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Oral tablets in 0.5mg or 0.75mg strength
  Other Names: Ondansetron HCl
  Arms: Ondansetron 0.5 mg; Ondansetron 0.75 mg
Drug: Placebo — Oral tablet to match the experimental interventions
  Arms: Placebo

SUMMARY:
This study is to assess the efficacy and safety of two doses of ondansetron (0.5 mg and 0.75 mg) relative to placebo when administered twice daily as adjunctive therapy for adult patients with Obsessive-Compulsive Disorder (OCD) who have not adequately responded to treatment with a serotonin reuptake inhibitor (SRI).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel-group study.

A sufficient number of patients will be screened to obtain approximately 150 patients randomized to the double-blind portion of the study. This study will consist of at least 6 weeks of retrospectively documented SRI treatment (prior to screening), 6 weeks of prospective SRI treatment after screening (run-in) but prior to randomization, and 12 weeks of double-blind treatment with study drug (ondansetron 0.5 mg twice a day, ondansetron 0.75 mg twice a day or placebo twice a day).

All patients will have been maintained on a single SRI at the same dose throughout the retrospective 6-week period and will continue the same SRI at the same dose throughout the run-in and double-blind treatment periods.

The 12-week randomized, double-blind, placebo-controlled, parallel-group study will be the "core period" for purposes of efficacy and short-term safety assessment. Patients completing all 12 weeks of the core period will be offered an opportunity to participate in an "extension period" where they will continue to receive treatment for up to 30 months following the core period.

Treatment assignment in the extension period will be as follows: responders will continue on the same double-blind treatment to which they were assigned in the core period (ondansetron 0.5 mg twice a day, ondansetron 0.75 mg twice a day, or placebo twice a day); non-responders will be reassigned to continuing treatment according to their prior treatment assignment in the core period (those who received placebo will be assigned to ondansetron 0.5 mg twice a day, those who received ondansetron 0.5 mg twice a day will be assigned to ondansetron 0.75 mg twice a day, and those who received ondansetron 0.75 mg twice a day will continue receiving ondansetron 0.75 mg twice a day). Patients will receive treatment under double-blind conditions (double-blind phase of the extension study) until the core study is completed and the safety and efficacy of an ondansetron dose has been confirmed

If after the core study data analysis, no treatment differences are found between ondansetron and placebo in the primary efficacy variable, the extension study will be terminated. If the core study results are positive for the primary efficacy endpoint and safety endpoints, then patients participating in the double-blind phase of the extension study will be offered an opportunity to continue treatment under open-label conditions with the dose deemed efficacious and safe (open-label phase of the extension study). A Data Review Committee will be responsible for reviewing the core study analysis results, providing a dose recommendation for the open-label phase of the extension study, and for communicating the results and their recommendation to the participating institutional review boards/ethics committees (IRBs/ECs) and investigators. Patients may continue receiving treatment for up to 30 months or until the sponsor provides an alternative.

ELIGIBILITY:
Core period: Inclusion criteria for entry in prospective serotonin reuptake inhibitor (SRI) period (screening):

* Male or female adults 18 years of age or older
* Able to understand the study and provide informed consent
* Subjects who are fluent in English and/or Spanish (speaking, writing, and reading)
* Willing and able to comply with the requirements of the protocol and follow directions from the clinic staff
* Body mass index (BMI) ≤ 40 kg/m^2 (wearing indoor clothing without shoes)
* For all females: Female patients will be included if they are post-menopausal for at least two years or sterilized, or if they are of childbearing potential, they are not breastfeeding, their pregnancy test is negative, they have no intention of becoming pregnant during the course of the study, and are using adequate contraceptive drugs or devices. Medically acceptable methods of contraception that may be used by the patient and/or her partner are: oral contraceptives, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization or abstinence. Females using oral contraception must have started using the medication at least 8 weeks prior to screening. Surgical sterilization must have occurred at least 6 weeks prior to screening.
* Documented diagnosis of Obsessive-Compulsive Disorder (OCD) as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria
* At screening, documented history of stable and current regimen of one of the following five serotonin reuptake inhibitor (SRI) for at least 6 weeks prior to screening at the minimum daily dosage listed:

  * clomipramine (Anafranil®) 150 mg
  * fluvoxamine (Luvox®) 200 mg or fluvoxamine CR (Luvox CR®) 200 mg
  * fluoxetine (Prozac®) 40 mg
  * paroxetine (Paxil®) 40 mg (does not include paroxetine CR (Paxil CR®))
  * sertraline (Zoloft®) 100 mg
* Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score of ≥ 24
* Hamilton Depression Rating Scale (HAM-D) score of < 20

Inclusion criteria for randomization to double-blind treatment period:

* During run-in, documented use of stable and current regimen of one of the following five serotonin reuptake inhibitor (SRI) for at least 6 weeks prior to screening at the minimum daily dosage listed:

  * clomipramine (Anafranil®) 150 mg
  * fluvoxamine (Luvox®) 200 mg or fluvoxamine CR (Luvox CR®) 200 mg
  * fluoxetine (Prozac®) 40 mg
  * paroxetine (Paxil®) 40 mg (does not include paroxetine CR (Paxil CR®))
  * sertraline (Zoloft®) 100 mg
* Demonstrated failure to adequately respond to serotonin reuptake inhibitor (SRI) treatment, defined by the following 2 criteria after 6 weeks of prospective treatment:

  * Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score ≥ 21
  * Less than 25% improvement in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score from Week -6 (screening)
* Hamilton Depression Rating Scale (HAM-D) score of ≤ 16

Extension Period - Inclusion criteria for randomization to double-blind extension treatment period:

* Completing 12 weeks of treatment in the double-blind core period
* Demonstrating compliance in the judgment of the investigator, with both the SRI and study drug as prescribed.

Core Period Exclusion Criteria:

* Presence of significant medical illnesses such as, but not restricted to, cardiovascular, (including congestive heart failure and bradyarrhythmias), endocrine or intestinal disorders that would interfere with the conduct of the study
* History of significant head injury, other significant brain trauma, or seizure disorder (not including a single childhood febrile seizure)
* Clinically significant abnormal laboratory findings. Presence of clinically significant electrolyte abnormalities will be exclusionary.
* Clinically significant abnormal findings on electrocardiogram (ECG). Diagnosis of congenital long QT syndrome will be exclusionary.
* Clinically significant abnormal findings on physical examination
* Positive pregnancy test
* Subjects who intend to donate blood or blood components while receiving study drug or within 1 month of the completion of treatment
* Hoarding as the primary Obsessive-Compulsive Disorder (OCD) symptom (secondary hoarding will be allowed)
* Obsessive-compulsive spectrum disorder as a primary disorder (secondary obsessive-compulsive spectrum disorders will be allowed)
* Requiring active behavioral therapy during the study period (run-in and treatment periods). Patients with a history of behavioral therapy may be enrolled as long as they will not be actively engaged in behavioral therapy during the study. However, booster sessions, occurring no more than quarterly (before and after the core study), are allowed. Supportive and other forms of psychotherapy will be permitted during the study as long as the patient has been engaged in such therapy for at least 8 weeks prior to study enrollment and there are no changes during the study.
* A history of substance dependence or drug or substance abuse, including alcohol abuse, within the past 12 months. A history of nicotine dependence will not be considered an exclusion criterion.
* Mental retardation or an IQ less than 70
* The following comorbid psychiatric conditions identified by current or past medical history or as a result of the Mini-International Neuropsychiatric Interview (MINI) or Structured Clinical Interview for DSM-IV-TR Axis II Personality Disorders (SCID-II) psychiatric interviews will be excluded:

  * Schizophrenia or other psychotic disorders
  * Schizotypal personality disorder
  * Bipolar disorder
  * Gilles de la Tourette syndrome
  * Autism and autistic spectrum disorders
  * Eating disorders
  * Combat-related post-traumatic stress disorder
  * Other comorbid anxiety disorders will be permitted if the severity will not interfere with study participation.
* Subjects who are believed to have suicidal or homicidal risk (i.e., after an assessment by a qualified mental health professional if the C-SSRS screening assessment warranted a suicidal risk assessment interview), or with a history of suicidality in the previous 3 months
* Taking trazodone or other medicinal products that have been associated with prolongation of the QT/QTc interval.
* Taking concomitant antipsychotic drugs, lithium, carbamazepine, oxcarbazepine, phenytoin, anti-anxiety drugs (other than the current SRI for treatment of OCD), or benzodiazepines prescribed for the treatment of anxiety. PRN use of FDA-approved benzodiazepine or non-benzodiazepine hypnotics will be allowed. In addition, the following 3 benzodiazepines will be allowed, provided that patients have been taking them only at bedtime as a sleep aid for at least 12 weeks at the maximum doses noted below:

  * clonazepam (Klonopin®) up to 1 mg
  * diazepam (Valium®) up to 5 mg
  * lorazepam (Ativan®) up to 1 mg
* Taking more than one SRI at the time of screening or at any time in the previous 8 weeks
* A history of having failed more than 2 prior treatments, not including their current course of treatment, with serotonin reuptake inhibitors (SRIs), including clomipramine and selective serotonin reuptake inhibitors (SSRIs), or serotonin-norepinephrine reuptake inhibitors (SNRIs) may only be considered after consultation with the medical monitor. Failure is defined as inadequate response, in the judgment of the treating physician, to an adequate dose of SRIs or SNRIs taken for at least 8 weeks.
* Taking any antidepressant drugs (including St. John's Wort), at the time of screening or at any time in the previous 8 weeks, other than the SRI identified in the retrospective and screening periods
* Likely to use triptans at any time during the run-in or double-blind portion of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Core Period: Change from baseline in the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) total at Month 3 score | Day -1 (baseline), Month 3
Extension Period: Participants with Safety Adverse Experiences | up to Month 33

SECONDARY OUTCOMES:
Core Period: Participants Considered Responders as Measured by the Clinical Global Impression-Improvement (CGI-I) Score | Month 3
Core Period: Change from Baseline in the Clinical Global Impression-Severity (CGI-S) Score at Month 3 | Day -1 (baseline), Month 3
Core Period: Change from Baseline in the Sheehan Disability Scale (SDS) Score at Month 3 | Day -1 (baseline), Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Study Chair — Montefiore Medical Center, Bronx, NY
Locations (32):
- United States (22):
  - Southwestern Research, Inc., Beverly Hills, California
  - Sun Valley Research Center, Imperial, California
  - Pacific Institute for Medical Research, Los Angeles, California
  - Compass Research, LLC, Orlando, Florida
  - University of South Florida, St. Petersburg, Florida
  - Emory University, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - McLean Hospital, Belmont, Massachusetts
  - Beacon Clinical Research, LLC, New Bedford, Massachusetts
  - Ambulatory Research Center, Dept of Psychiatry, Minneapolis, Minnesota
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Biobehavioral Institute, Hofstra, Great Neck, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Columbia University Medical Center NYS Psychiatric Institute, New York, New York
  - Montefiore Medical Center, Child Psychiatry Annex, The Bronx, New York
  - Richard H. Weisler, MD, PA, and Associates, Raleigh, North Carolina
  - Quest Therapeutics of Avon Lake, Avon Lake, Ohio
  - Lindner Center of HOPE University of Cincinnati, Mason, Ohio
  - The Body Dysmorphic Disorder (BDD) Program, Providence, Rhode Island
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Dean Foundation, Middleton, Wisconsin
  - The Rogers Center for Research and Training, Milwaukee, Wisconsin
- Mexico (10):
  - Grupo de Estudios Medicos y Familiares, Mexico City, Federal District
  - Instituto Mexicano de Investigacion Clinica S.A. de C.V. (IMIC), Mexico City, Federal District
  - Hospital Aranda de la Parra S.A. de C.V., León, Guanajuato
  - Estudios Integrales en Salud Mental, S.C., Guadalajara, Jalisco
  - CIT Neuropsique, Monterrey, Nuevo León
  - Centro par alas Adicciones y Salud Mental S.A., Monterrey, Nuevo León
  - Instituto de Informacion e Investigacion en Salud Mental, A.C. (INFOSAME), Monterrey, Nuevo León
  - Hospital Lomas de San Luis Internacional, San Luis Potosí City, San Luis Potosí
  - Instituto para el Fortalecimiento de Capacidades en Salud, Tlalnepantla, State of Mexico
  - Instituto para el Fortalecimiento de Capacidades en Salud: Focus Salud Mexico S.C., Mérida, Yucatán